CLINICAL TRIAL: NCT07297875
Title: A Phase Ⅰ/Ⅱ, Open-Label Study of ABSK061 to Assess Safety, Tolerability, Pharmacokinetics, and Efficacy in Children With Achondroplasia
Brief Title: A Study of ABSK061 to Assess Safety, Tolerability, Pharmacokinetics, and Efficacy in Children With Achondroplasia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK061-202
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABSK061 (Experimental): Dose escalation part will be divided into Part A and Part B according to patient age, with Part A enrolling children with ACH aged 6 to < 12 years (inclusive of 6 years) and Part B enrolling children with ACH aged 3 to < 6 years (inclusive of 3 years). In this study, two sentinel patients will be set for both parts of each dose level, thereby the interval for the first dose between the first 2 patients and the third patient is not less than 28 days.
  This study will employ the Bayesian optimal interval (BOIN) design for dose escalation part to guide dose escalation. The target toxicity rate for the MTD is φ = 0.25 and the maximum sample size for the dose escalation part will be 80 (50 in Part A and 30 in Part B). The DLT observation period is defined as the first 28 days after administration of ABSK061.
  After the RDE is confirmed in the dose Escalation part, the dose Expansion phase will be conducted.
  Interventions: Drug: ABSK061

INTERVENTIONS:
Drug: ABSK061 — ABSK061 is supplied as minitablets filled in capsules. Four strengths of capsules will be provided: 0.2 mg, 2 mg, 3 mg, and 5 mg. Each patient can only be administered with a single strength.
  All patients will be administered orally once daily under the fasted state, i.e., fast from 2 hours before dosing to 1 hour after dosing. Dose will be calculated based on the patient's weight, and detailed rules for dose calculation are provided.
  Take out the ABSK061 capsule containing minitablets, take off the capsule cap and decant the content (minitablets), swallow the minitablets completely with water without chewing (the recommended water volume is 50-180 mL). If there is difficulty swallowing all the minitablets at once, they may be taken in several portions as needed, but the entire dose should be taken within 10 minutes. If needed, yogurt or apple sauce can be used as vehicles to facilitate swallowing of the minitablets.

SUMMARY:
This is a multicenter, non-randomized, open-label, phase I/II study in children with ACH. This study will start with a dose escalation of ABSK061 in children with ACH to evaluate the safety, tolerability, PK, and efficacy. The RDE confirmation part will evaluate the safety and efficacy of ABSK061 at the recommended doses for expansion (RDEs) in children with ACH. All patients enrolled in the dose escalation part and RDE confirmation part can enter the extended treatment period to further evaluate the long-term safety, tolerability, and long-term efficacy of ABSK061 in children with ACH.

DETAILED DESCRIPTION:
Up to 50 children aged 6 to < 12 years (inclusive of 6 years) with ACH and up to 30 children aged 3 to < 6 years (inclusive of 3 years) with ACH are expected to be enrolled in the dose escalation part of the study; up to 30 children aged 3 to < 12 years (inclusive of 3 years) with ACH are expected to be enrolled in the RDE confirmation part.

Children enrolled in this study will be required to complete at least 6 months and up to 2 years of growth assessment and observation of natural history of ACH in the sponsor's observational study (ABSK061-001).

Dose Escalation Part All patients enrolled in the dose escalation part will continue to receive ABSK061 once daily (QD) dosing frequency and will enter the extended treatment period for 52 weeks after completing 26 weeks of treatment.

The dose escalation includes a total of 5 potential dose levels starting at an initial dose of 0.064 mg/kg QD. In the absence of DLTs or ≥ grade 2 drug-related adverse events, the initial maximum permitted dose increment will not exceed 200%. In the presence of a DLT or ≥ grade 2 drug-related adverse event, dose escalation for subsequent cohorts will follow a modified Fibonacci scheme, in which the first two consecutive dose cohorts will each receive a maximum dose increase of up to 67% and 50%, respectively, and the remaining dose cohorts will receive a maximum of 33% increase. The potential dose levels to be explored are listed in the table below. Based on cumulative safety, PK/PD, efficacy data, other potential dose levels not listed may also be explored in this study following the dose escalation rules.

Dose escalation part will be divided into Part A and Part B according to patient age, with Part A enrolling children with ACH aged 6 to < 12 years (inclusive of 6 years) and Part B enrolling children with ACH aged 3 to < 6 years (inclusive of 3 years). In this study, two sentinel patients will be set for both parts of each dose level, thereby the interval for the first dose between the first 2 patients and the third patient is not less than 28 days.

RDE Confirmation Part In this part, up to 30 children aged 3 to < 12 years (inclusive of age 3) with ACH will be enrolled to receive one or two RDEs. The RDEs will be selected from the safe doses determined in the dose escalation to further evaluate the safety and efficacy of ABSK061 in children with ACH. Patients in this part will not be included in the DLT evaluable population. Dose decisions for RDE Confirmation Part will be based on discussion and alignment between the sponsor and investigators. Safety, PK/PD, and efficacy data will be monitored and assessed in real time during the study. The study may be discontinued early if any safety risk to the patients are identified, upon agreement between the investigators and sponsor.

Extended Treatment Period After completing 26 weeks of treatment with ABSK061 in the dose escalation part and RDE confirmation part, children with ACH will enter the extended treatment period for 52 weeks to further assess the long-term safety, tolerability and efficacy. In extended treatment period, patients will be treated at the dose assigned for dose escalation (intra-patient dose escalations are allowed for patients at low dose levels in Part A). Dose will be calculated based on body weight and may be adjusted due to weight change at the Week 27 (W27D1, i.e., just entering the extended treatment period), Week 41 (W41D1), Week 53 (W53D1), and Week 67 (W67D1) visits.

After completing 78 weeks of study treatment set in the protocol, all patients in this study can be enrolled into a separate long-term extension study conducted by the sponsor to continue ABSK061 treatment. This is to further assess the long-term safety and efficacy of ABSK061 in children with ACH. If the investigator determines that a patient is no longer eligible to continue in the long-term extension study due to safety concerns or lack of clinical benefit, treatment with ABSK061 will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to screening, the guardians and children with ACH (if applicable) must voluntarily provide signed informed consent.
2. Patients with a clear clinical diagnosis of ACH confirmed by genetic testing for an FGFR3 mutation.
3. Male or female, age at screening:

   Dose Escalation Part A: 6 to < 12 years (inclusive 6 years) Dose Escalation Part B: 3 to < 6 years (inclusive 3 years) RDE Confirmation Part: 3 to < 12 years (inclusive 3 years).
4. Have completed at least 6 months (i.e., the "Day 181" visit) of growth assessment and observation of natural history of ACH in the observational study (ABSK061-001) before study entry.
5. Tanner Stage 1 breast development for females or Tanner Stage 1 external genitalia development for males at screening

Exclusion Criteria:

1. Known allergy or hypersensitivity to any component of the study drug.
2. Bone age ≥ 14 years as assessed by the investigator based on hand and wrist X-ray.
3. Have a form of skeletal dysplasia other than ACH or known medical conditions that result in short stature or abnormal growth, including but not limited to severe achondroplasia with developmental delay and acanthosis nigricans (SADDAN), Turner syndrome, pseudoachondroplasia, inflammatory bowel disease, chronic renal insufficiency, active celiac disease a, Vitamin D deficiency b, untreated hypothyroidism c, poorly controlled diabetes (HbA1c ≥8.0%) or diabetic complications
4. History or presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones.
5. AGV ≤ 1.5 cm/year over at least 6 months (i.e., must have completed the 'Day 181' visit) in the observational study (ABSK061-001), or current evidence of growth plate closure (proximal tibia, distal femur).
6. Current epiphyseal injury (Salter-Harris fracture) or severe hip pain.
7. For ACH-related complications: current severe sleep apnea, symptomatic and/or requiring intervention for hydrocephalus, or spinal cord compression at the cranio-cervical junction, or prior ventriculoperitoneal shunt surgery.
8. Have received any dose of medications affecting stature or body proportionality, such as human growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids within 12 months prior to screening.
9. Prior treatment with any CNP analogues or FGFR inhibitors. Prior use of any investigational drugs or investigational medical devices that affect height or body proportion.
10. History of any prior bone-related surgery that affects long bone growth, such as orthopaedic reconstructive surgery, limb lengthening, or osteotomy (patients who have previously undergone foramen magnum decompression or intervertebral disc/laminectomy are allowed if they have fully recovered after surgery and bone healing has occurred for at least 6 months. Patients who have previously undergone eight-plate epiphysiodesis are allowed if the plate has been removed and healed for at least 4 weeks).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2031-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Day 1 to Day 28 of dosing
  Incidence of dose-limiting toxicities (DLTs) in the DLT observation period, defined as Day 1 to Day 28 of dosing
Incidence and severity of adverse events (AEs) | up to 87 weeks
  Incidence and severity of adverse events (AEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) using Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0), and relatedness, rate of dose modifications (including dose interruption and dose reduction) or discontinuation of study drug due to toxicity, and changes from baseline in safety assessments such as laboratory parameters, x-ray, electrocardiograms (ECGs), echocardiograms, vital signs, and physical examinations (including ophthalmic examinations)
Changes from baseline in the Annualized Growth Velocity (AGV, cm/year) | Day 1 of dosing to 78-week End of Treatment
  Changes from baseline in the Annualized Growth Velocity (AGV, cm/year) over 52 weeks [baseline is defined as the AGV obtained through at least 6 months of observation in the observational study (ABSK061-001)]

SECONDARY OUTCOMES:
Cmax | Day 1 of dosing to 78-week End of Treatment
  maximum observed concentration
Tmax | Day 1 of dosing to 78-week End of Treatment
  time to maximum observed concentration
AUC | Day 1 of dosing to 78-week End of Treatment
  area under the concentration-time curve
t1/2 | Day 1 of dosing to 78-week End of Treatment
  half-life
Vz/F | Day 1 of dosing to 78-week End of Treatment
  apparent volume of distribution
CL/F | Day 1 of dosing to 78-week End of Treatment
  apparent oral clearance
Cmax,ss | Day 1 of dosing to 78-week End of Treatment
  maximum observed concentration of steady/state
Cmin,ss | Day 1 of dosing to 78-week End of Treatment
  minimum observed concentration of steady/state
AUCtau,ss | Day 1 of dosing to 78-week End of Treatment
  area under the concentration-time curve after multiple dose
AR | Day 1 of dosing to 78-week End of Treatment
  accumulation ratio
standing height | Day 1 of dosing to 78-week End of Treatment
  calculated to the nearest 0.1 cm
sitting height | Day 1 of dosing to 78-week End of Treatment
  calculated to the nearest 0.1 cm
sitting height to standing height ratio | Day 1 of dosing to 78-week End of Treatment
  This parameter is calculated as the ratio of sitting height to total standing height. It is used to assess the abnormality in body proportions, specifically the relative trunk-to-lower limb length. In patients with achondroplasia, this ratio is typically increased. Within the clinical trial, this measure is used to evaluate the treatment drug's effect on body proportions.
height Z scores | Day 1 of dosing to 78-week End of Treatment
  This measure is defined as the number of standard deviation units by which the subject's height differs from the mean height of a healthy, age- and sex-matched reference population. It is a standardized value used to precisely quantify the degree of deviation from the normal growth curve. In the clinical trial, it serves as a key parameter for assessing the treatment's efficacy in improving linear height growth.

OTHER OUTCOMES:
Range of Motion (ROM) | Day 1 of dosing to 78-week End of Treatment
  Mean change from baseline in ROM of the affected joint

CONTACTS AND LOCATIONS:
Overall Officials: Shuqi Zeng, Study Director — 12B, Building 1, No 515, Huanke Road, Pudong New Area, Shanghai 201210, China
Locations (7):
- China (7):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Henan Children's Hospital, Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengde, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No